CLINICAL TRIAL: NCT05370898
Title: Clinical Study of Bugu Shengsui Decoction for the Treatment of Primary Osteoporosis (Kidney Yang Deficiency Syndrome)
Brief Title: The Study of Chinese Medicine for the Treatment of Primary Osteoporosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wangjing Hospital, China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZZ13-YQ-039
Record Dates: First submitted 2022-04-13; First posted 2022-05-12 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Primary Osteoporosis
Keywords: Traditional Chinese medicine intervention; Completely randomized controlled trial; Double blind method clinical trial; Efficacy evaluation; Mechanism research

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Chinese medicine (Experimental): On the basis of general symptomatic treatment of caltrate D，patients in experimental group use the traditional Chinese medicine application prescription.
  Interventions: Drug: Caltrate D; Drug: Chinese medicine prescription
- Comparator: placebo (Placebo Comparator): On the basis of general symptomatic treatment of caltrate D，patients in placebo group use the simulate granule of traditional Chinese medicine application prescription.
  Interventions: Drug: Caltrate D; Drug: Placebo

INTERVENTIONS:
Drug: Caltrate D — Caltrate D is allowed for basic treatment when the patient is diagnosed with primary osteoporosis (Kidney Yang Deficiency Syndrome).Take it continuously for 3 months.
Drug: Chinese medicine prescription — The Chinese medicine application prescription is composed of Rhizoma Drynariae 12g, psoralen 10g, dog ridge 10g, medlar 10g, raw oyster 10g, ginseng 6g, Panax notoginseng 3g, Amomum villosum 6g.Patients take 200ml each time, twice a day. Treatment duration are 3 months.
  Arms: Traditional Chinese medicine
Drug: Placebo — The placebo is simulate granule of Chinese medicine application prescription. Patients take 200ml each time, twice a day. Treatment duration are 3 months.
  Arms: Comparator: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and possible mechanism of traditional Chinese medicine in the treatment of primary osteoporosis (Kidney Yang Deficiency Syndrome).It is a randomized, placebo-controlled trial.

DETAILED DESCRIPTION:
The subjects are selected according to the inclusion criteria and exclusion criteria. Using the network random system, 120 subjects who meet the research criteria are randomly divided into control group and experimental group, with 60 cases in each group. Patients in treatment group take the granule of traditional Chinese medicine prescription, while the control group take simulate granule of the prescription. Both two groups are under symptomatic treatment. Twice a day, in the morning and evening, 30 minutes after meals.The experimental drugs were provided by the pharmacy department of Wangjing hospital, Chinese Academy of traditional Chinese medicine, and the course of treatment was 3 months.The observation time points were before treatment, 2 weeks after treatment, 1 month after treatment and 3 months after treatment. Visual Analogue Score (VAS), Traditional Chinese Medicine（TCM）syndrome score, SF-12 scale and bone metabolism index were used as observation indexes.At the same time, it is planned to determine EphrinB2, EphB4, Runx2 and VEGF in serum by ELISA.

Tele-medicine and information management system is established to help achieve follow-up interviews.Random numbers are generated by SAS 9.4 software. The subjects, caregivers, investigators and outcomes assessors in this study are all blinded.

ELIGIBILITY:
Inclusion Criteria:

1. It meets the diagnostic criteria of Western medicine for primary osteoporosis. the diagnostic criteria of osteoporosis based on the bone mineral density of central axis (lumbar spine 1-4, femoral neck or total hip) or 1/3 bone mineral density of distal radius measured by DXA is t-value ≤ - 2.5;
2. It meets the syndrome differentiation standard of primary osteoporosis with Kidney Yang Deficiency Syndrome;
3. Female menopause > 2 years and 45 years ≤ age < 80 years, or 50 years ≤ male < 80 years;
4. Visual Analogue Score (VAS) was used to evaluate pain ≥ 4 points;
5. Voluntarily participate in this clinical study and sign the informed consent form.

Exclusion Criteria:

1. Osteoporotic fracture has occurred, or t-value > - 2.5;
2. Female premenopausal or menopausal years ≤ 2 years, female age < 45 years or ≥ 80 years, male age < 50 years or ≥ 80 years;
3. VAS pain score < 4;
4. Lumbar fusion or severe degenerative changes hinder the measurement of normal bone mineral density, and there are less than 2 consecutive intact lumbar vertebrae for DXA measurement and evaluation;
5. Patients with malignant tumor, cardiovascular, cerebrovascular, liver disease, kidney disease, hematopoietic system and other serious primary diseases;
6. secondary osteoporosis: diabetes, thyroid disease, Cushing syndrome and other metabolic diseases, rheumatoid arthritis, multiple myeloma, gout, absorption syndrome, systemic lupus erythematosus and other systemic diseases.
7. Use drugs affecting bone metabolism, such as bisphosphonates, glucocorticoids, calcitonin, anticonvulsant drugs, heparin and other drugs within 3 months before signing the informed consent;
8. History of serious mental illness or poor compliance;
9. Allergic constitution, allergy to known components of the drug, allergy to calcium or vitamin D;
10. Those who participated in other clinical trials within 3 months.

Rejection Criteria:

1. False diagnosis and false inclusion;
2. Not receiving one treatment;
3. During the study, in addition to the study medication, drugs known or likely to affect bone metabolism were used.

Shedding Standard:

1. The subjects withdrew from the test by themselves;
2. Loss of follow-up;
3. The subject received treatment at least once, and there were serious complications or complications and serious adverse events;
4. Although the test was completed, the dosage of the subject was not within the range of 80%-120% of the dosage that should be taken.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female：menopause > 2 years and 45 years ≤ age < 80 years Male：50 years ≤ male < 80 years;
Enrollment: 120 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Change of VAS pain score of low back | Change from baseline VAS score at 2 weeks.
  Draw a straight line with a length of 10 cm on the white paper and mark "painless" and "severe pain" on both ends respectively to form VAS. The patient makes a mark on the straight line according to the degree of pain he feels. The distance from the starting point to the mark is the quantified degree of pain. Painless is represented by 0; 1-3 points represent mild pain; 4-6 points represent moderate pain, which is strong but tolerable; 7-10 points represent severe pain, gradually reaching intolerable level, which is severe pain.
Change of VAS pain score of low back | Change from baseline VAS score at 1 month.
  Draw a straight line with a length of 10 cm on the white paper and mark "painless" and "severe pain" on both ends respectively to form VAS. The patient makes a mark on the straight line according to the degree of pain he feels. The distance from the starting point to the mark is the quantified degree of pain. Painless is represented by 0; 1-3 points represent mild pain; 4-6 points represent moderate pain, which is strong but tolerable; 7-10 points represent severe pain, gradually reaching intolerable level, which is severe pain.
Change of VAS pain score of low back | Change from baseline VAS score at 3 months.
  Draw a straight line with a length of 10 cm on the white paper and mark "painless" and "severe pain" on both ends respectively to form VAS. The patient makes a mark on the straight line according to the degree of pain he feels. The distance from the starting point to the mark is the quantified degree of pain. Painless is represented by 0; 1-3 points represent mild pain; 4-6 points represent moderate pain, which is strong but tolerable; 7-10 points represent severe pain, gradually reaching intolerable level, which is severe pain.
Change of Traditional Chinese medicine (TCM) syndrome score | Change from baseline TCM syndrome score at 2 weeks.
  According to the《expert consensus on the prevention and treatment of primary osteoporosis with reference to traditional Chinese medicine (2020)》, the quantitative evaluation table of TCM syndrome differentiation for osteoporosis with Kidney Yang Deficiency syndrome was formulated to evaluate the symptoms. Symptoms include primary and secondary symptoms, the primary symptoms were low back pain and soreness and weakness, the secondary symptoms include restricted movement of the lumbar spine，fear of cold and like to be warm，degree of frequency of urination. The primary symptom score was 0 (absent), 2 (mild), 4 (moderate), or 6 (marked)，the secondary symptom score was 0 (absent), 1 (mild), 2 (moderate), or 3 (marked).The obtained scores were summed to calculate the total score.
Change of Traditional Chinese medicine (TCM) syndrome score | Change from baseline TCM syndrome score at 1 month.
  According to the《expert consensus on the prevention and treatment of primary osteoporosis with reference to traditional Chinese medicine (2020)》, the quantitative evaluation table of TCM syndrome differentiation for osteoporosis with Kidney Yang Deficiency syndrome was formulated to evaluate the symptoms. Symptoms include primary and secondary symptoms, the primary symptoms were low back pain and soreness and weakness, the secondary symptoms include restricted movement of the lumbar spine，fear of cold and like to be warm，degree of frequency of urination. The primary symptom score was 0 (absent), 2 (mild), 4 (moderate), or 6 (marked)，the secondary symptom score was 0 (absent), 1 (mild), 2 (moderate), or 3 (marked).The obtained scores were summed to calculate the total score.
Change of Traditional Chinese medicine (TCM) syndrome score | Change from baseline TCM syndrome score at 3 months.
  According to the《expert consensus on the prevention and treatment of primary osteoporosis with reference to traditional Chinese medicine (2020)》, the quantitative evaluation table of TCM syndrome differentiation for osteoporosis with Kidney Yang Deficiency syndrome was formulated to evaluate the symptoms. Symptoms include primary and secondary symptoms, the primary symptoms were low back pain and soreness and weakness, the secondary symptoms include restricted movement of the lumbar spine，fear of cold and like to be warm，degree of frequency of urination. The primary symptom score was 0 (absent), 2 (mild), 4 (moderate), or 6 (marked)，the secondary symptom score was 0 (absent), 1 (mild), 2 (moderate), or 3 (marked).The obtained scores were summed to calculate the total score.
Change of 12-Item Short Form Survey (SF-12) score | Change from baseline SF-12 score at 1 month.
  The 12-Item Short Form Survey have 12 items and 8 dimensions, which are overall health, Physical Functioning, Role-Physical, Bodily Pain, Vitality, Social Functioning, Role-Emotional and Mental Health. The first four dimensions belong to the level of Physical Component Summary, and the last four dimensions belong to the level of Mental Component Summary. Each item was scored according to the corresponding options to evaluate the impact of health on an individual's everyday life. The highest score of item 2 and 3 is 3, and the lowest score is 1. The highest score of the other ten items is 5, and the lowest score is 1. The obtained scores were summed to calculate the total score to evaluate the changes of patients' quality of life.The higher the score, the better the quality of life.
Change of 12-Item Short Form Survey (SF-12) score | Change from baseline SF-12 score at 3 months.
  The 12-Item Short Form Survey have 12 items and 8 dimensions, which are overall health, Physical Functioning, Role-Physical, Bodily Pain, Vitality, Social Functioning, Role-Emotional and Mental Health. The first four dimensions belong to the level of Physical Component Summary, and the last four dimensions belong to the level of Mental Component Summary. Each item was scored according to the corresponding options to evaluate the impact of health on an individual's everyday life. The highest score of item 2 and 3 is 3, and the lowest score is 1. The highest score of the other ten items is 5, and the lowest score is 1. The obtained scores were summed to calculate the total score to evaluate the changes of patients' quality of life.The higher the score, the better the quality of life.
Changes of serum bone metabolic indexes | Change from baseline bone metabolism index at 3 months.
  Serum level of Beta-CrossLaps (β-CTX) in ng/mL, N-terminal propeptide of type I procollagen (P1NP) in ng/mL，which are determined by Electrochemiluminescence Method.The normal reference ranges of serum P1NP and β-CTX are 16.3~78.2 ng/mL and 0.114~0.628ng/mL, respectively.In case of abnormal conditions,the higher the β-CTX, the more serious the bone resorption.The lower the P1NP, the less bone formation and the worse the bone condition.
Changes of serum ALP | Change from baseline ALP at 3 months.
  Serum level of Alkaline phosphatase (ALP) in U/L, which is determined by automatic biochemical analysis.The normal value is 40-150 U/L.When it is lower than the normal value, it indicates that bone formation is reduced.
Changes of serum BGP | Change from baseline BGP at 3 months.
  Serum level of bone glaprotein (BGP) in μg/L, which is determined by automatic biochemical analysis.The normal value is 4.8~10.2 μg/L.When it is lower than the normal value, it indicates that bone formation is reduced.
Changes of serum 25OHD | Change from baseline 25OHD at 3 months.
  Serum level of 25-hydroxy vitamin D (25OHD) in nmol/ml，which is determined by Electrochemiluminescence Method. Its value ≥ 30 nmol/L is normal，it may appear osteoporosis if below this value.

SECONDARY OUTCOMES:
Therapeutic mechanism | Change from baseline at 3 months.
  Serum level of EphrinB2, EphB4, Runx2 and VEGF in μg/mL，which is determined by enzyme linked immunosorbent assay（ELISA）.The higher the value, the better the bone condition. So as to verify the mechanism of Bugu Shengsui decoction.

OTHER OUTCOMES:
Blood routine tests | Up to 3 months.
  Blood routine tests are performed with a blood routine analyzer to monitor the patient's health status.A normal blood routine indicates that the drug has no side effects. If abnormal conditions occur, take appropriate measures to treat them.
Electrocardiogram | Up to 3 months.
  Electrocardiogram（ECG） tests using an electrocardiograph to monitor the patient's health, a normal ECG indicates that the drug has no adverse effects. If abnormal conditions occur, appropriate measures should be taken to deal with them.
Blood urea nitrogen | Up to 3 months.
  Blood urea nitrogen（Bun）is detected by kinetic rate method to monitor the renal function of the patient, a normal Bun indicates that the drug has no adverse effects. Its normal value is 2.9～7.5 mmol/L. If abnormal conditions occur, appropriate measures should be taken to deal with them.
Serum creatinine | Up to 3 months.
  Serum creatinine (Cr) is detected by kinetic rate method to monitor the renal function of the patient, a normal Cr indicates that the drug has no adverse effects. Its normal value is 44-133 μmol/L. If abnormal conditions occur, appropriate measures should be taken to deal with them.
Liver function | Up to 3 months.
  Alanine aminotransferase（ALT）、Aspartate aminotransferase（AST）、Gamma-glutamyltransferase（γ-GT） are detected by kinetic rate method to monitor the liver function of the patient, normal liver function indicate that the drug has no adverse effects. Their normal values are 0-40 U/L. If abnormal conditions occur, appropriate measures should be taken to deal with them.
Adverse events | Up to 3 months.
  umber of participants with treatment-related adverse events as assessed by CTCAE v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Wei, Ph.D, Study Director — Wangjing Hospital of China Academy of Chinese Medical Sciences; Ning Liu, Ph.D, Principal Investigator — Wangjing Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Wangjing Hospital of China Academy of Chinese Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided